CLINICAL TRIAL: NCT03322696
Title: STUDY OF THE ADAMTS-13 LEVEL AS PREDICTIVE BIOMARKER FOR DEVELOPMENT OF PORTAL VEIN THROMBOSIS IN LIVER CIRRHOSIS
Brief Title: ADAMTS-13 LEVEL AS PREDICTIVE BIOMARKER FOR DEVELOPMENT OF PORTAL VEIN THROMBOSIS IN LIVER CIRRHOSIS (ADAPTHRO)
Acronym: ADAPTHRO
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Raimondo De Cristofaro (Other)
Responsible Party: Sponsor-Investigator, Raimondo De Cristofaro, Prof. Raimondo De Cristofaro, MD, Catholic University of the Sacred Heart
Organization: Catholic University of the Sacred Heart (Other)
Other Study IDs: 0014168/17
Record Dates: First submitted 2017-10-23; First posted 2017-10-26 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Liver Cirrhosis
Keywords: ADAMTS-13, Liver Cirrhosis, Portal Vein Thrombosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cirr-PVT: Cirrhotic patients developing over 1 yr period thrombosis of portal vein or collaterals

SUMMARY:
Patients with cirrhosis of viral etiology (HCV/HBV); Patients with cirrhosis of any other etiology (alcohol, idiopatic, autoimmune). Planned Number of cirrhotic subjects 200 patients Inclusion Criteria Subjects (18 yr old) with liver cirrhosis of any etiology, Exclusion Criteria All patients should not have hepatocellular carcinoma or other malignant tumors, they should not be treated with anticoagulant / antiplatelet agents, not affected by PVT already diagnosed and not suffering from congenital coagulation disorders (haemophilia A / B, von disease Willebrand, another congenital deficiency of coagulation factors) or severe thrombocytopenia (<30,000 Plt / μL). Subject has participated in another clinical study within 30 days prior to study enrollment or is scheduled to participate in another clinical study on cirrhosis Primary Objective To describe the prospective modification of ADAMTS-13 level and other coagulation variables (e.g. FVIII, VWF:Ag/VWF:act) in cirrhotic patients during 18 months from the enrolment and to verify their predictive role as biomarker of development of portal vein thrombosis (PVT) Secondary Objectives To describe prospectively the modification of ADAMTS-13 level as a function of the etiology of cirrhosis Statistical analysis The total duration of the study will be of 12 months. The sample size of 200 subjects will be selected as a feasible number of patients to be recruited in a period of six months. The patients will be consecutively enrolled and followed for 18 months. As a result, in a follow up period of 18 months about 20-25 cases of PVT are expected. Continuous variables will be expressed as means ± standard deviations. In addition to descriptive statistics (location parameters), univariate analysis will be performed on each parameter and development of PVT during the follow up period. In previous observational studies both 1) a reduced PV flow [prospectively] and 2) a reduction of ADAMTS-13 are significantly associated with PVT. These associations will be investigated prospectively and analyzed simultaneously by a multivariate analysis and ROC curve to establish the sensitivity and specificity of these parameters as predictors of PVT development. Analyses will be performed using available data

DETAILED DESCRIPTION:
BACKGROUND AND JUSTIFICATION The occurrence of portal vein thrombosis (PVT) radically changes the prognosis of cirrhotic patients, particularly those awaiting liver transplantation. If this happens, it occurs in about 8-10% / year in patients with cirrhosis awaiting liver transplantation. Some studies have suggested the involvement of various risk factors for the development of PVT in cirrhotic patients, including the classic congenital and acquired thrombophilic conditions [1-6], although contributions of our research group have shown that a key element in the development of PVT in these patients is the decreased velocity of portal blood flow [7, 8]. The possible contribution of the von Willebrand factor (VWF) and ADAMTS-13, produced by the liver stellate cells [9], for the development of PVT is rather poorly documented. In a recent observational study of the proponent [10], conducted on 84 patients with liver cirrhosis, it was found that the level of circulating ADAMTS-13 is significantly lower in the group with PVT (median = 16.8% vs. 69.1%, p = 0.0047) and independently associated with the presence of portal thrombosis (p = 0.007). However, given the non-longitudinal nature of the study, it is possible that the decreased level of ADAMTS-13 observed is the consequence and not the cause of PVT. It is also yet to investigate the association of ADAMTS-13 level with the specific etiology of cirrhosis (viral, alcoholic, idiopathic, etc.) and the resulting inflammation during the course of the disease.

Duration of Study Period(s) and Subject Participation Two hundred (200) patients, consecutively enrolled in a period of about 6 months, will be followed for 18 months from the enrolment. As a result, in the subsequent 18 months about 20-25 cases of PVT will be expected. All patients will sign an informed consent. The severity of liver function failure will be assessed using the Child-Pugh score [11].

Primary Endpoint To describe in a prospective way the association of both basal ADAMTS-13 level and portal vein flow with development of PVT in cirrhotic patients during 18 months from the enrolment. Secondary Endpoints To describe prospectively the modification of ADAMTS-13 level as a function of the etiology of cirrhosis Coagulation and biochemical parameters

The prospective study will measure the following biochemical and coagulation parameters at each follow-up visit, scheduled at interval of 4 months according to routine controls:

Coagulation and thrombophilia factors All blood samples will be drawn under fasting conditions in the morning. Determinations of PT, APTT, fibrinogen, antithrombin, protein C, protein S, lupus anticoagulant, FVIII (two-stage chromogenic assay) and D-dimer will be carried out on an automatic coagulometer (ACL Top 700, IL). VWF-antigen VWF:activity will be measured in plasma samples by chemiluminescence assays. VWF multimer (VWFm) pattern was measured as previously reported [10]. FV Leiden R506Q and prothrombin G20210A genotyping of these polymorphisms was performed by using commercial kits based on PCR-RT-based method (from EliTechGroup S.p.A., Torino, Italy) on an automatic instrument (Model 7300, Applied Biosystem, Foster City, CA, USA).

Measurement of ADAMTS-13 activity. ADAMTS-13 activity was measured in citrated plasma samples by a fluorescence resonance energy transfer (FRET)-based assay using a VWF86 amino-acid peptide substrate contained in a commercial kit from Instrumentation Laboratory (ADAMTS-13 activity, Werfen Group, Milano, Italy) and a Varian Eclipse spectrofluorometer, as previously detailed [10, 13] and expressed as % of normal plasma.

Clinical Chemistry assays. All clinical chemistry assays (plasma albumin, creatinine, alanine-leucine-amino-transferase (ALT) and total bilirubin) will be performed as a part of routine diagnostic work-up within 24 hours of clinical observation in the central laboratory of the "A. Gemelli" Hospital, using heparinized plasma samples and commercial reagents from Siemens.

Secondary objectives. The secondary objectives of analyzing the levels of ADAMTS-13 and VWF as a function of the etiology of cirrhosis will be further assessed only after a certified diagnosis of the particular etiologic of cirrhosis. In the case of HCV-associated cirrhosis also the genotype of HCV will be analyzed.

Informed Consent and Enrollment Any patient who will provide informed consent (i.e., signs and dates the informed consent form and assent form, if applicable) and will meet all other inclusion/exclusion criteria will be considered enrolled in the study.

Subject Identification Code. The following series of numbers will comprise the subject identification code (SIC): protocol acronym (ADAPTHRO), and 2-digit subject number (e.g., 01….02) reflecting the order of enrollment (i.e., signing the informed consent form). For example, the third subject who signed an informed consent form will be identified as ADAPTHRO-03. All study documents (e.g., CRFs, clinical documentation, etc.) will be identified with the SIC.

Screening and Study Visits The study site is responsible for maintaining an enrollment/screening log that includes all subjects enrolled. The log also will serve to document the reason for screening failure. All screening data will be collected and reported in CRFs, regardless of screening outcome.

Subject Completion/Discontinuation A subject is considered to have completed the study when he/she ceases active participation in the study because the subject has, or is presumed to have, completed the study according to the protocol, participated for the specified observational time and when the study exit form has been completed. Reasons for completion/discontinuation will be reported on the Completion/ Discontinuation CRF page, including: completed, screen failure, adverse event (e.g., death), discontinuation by subject (e.g., lost to follow-up [defined as 3 documented unsuccessful attempts to contact the subject], dropout), physician decision (e.g., pregnancy, progressive disease, protocol violation(s)), Vital Signs Vital signs will include height (cm) and weight (kg). Height and weight will be collected, if available, at screening visit, each annual interval visit, and study completion/termination.

STATISTICAL ANALYSIS. Planned Statistical Analysis Continuous variables will be expressed as means ± standard deviations. Categorical variables will be expressed as frequencies and percentages. Fisher's exact tests and/or Chi-Square tests will be mainly used to compare qualitative variables and Student's t-test for quantitative unpaired data. A p-value < 0.05 will be considered statistically significant in an exploratory sense. In addition to descriptive statistics (location parameters), and univariate analysis, multivariate analyses are planned. Independent variables that will be found associated with PVT in univariate analysis with p<0.05 will be used as independent covariates associated with PVT in the next 18 months in the multivariable logistic regression analysis. A two-sided p <0.05 was defined as statistically significant. Analyses will be performed using SPSS software (version 21, Chicago, IL, USA) and GraphPad Prism software (GraphPad Software, Inc, La Jolla, CA, USA).

Informed Consent. Investigators will choose patients for enrollment based on the study eligibility criteria.The investigator will exercise no selectivity so that no bias is introduced from this source. All patients must sign an informed consent form before entering into the study according to applicable regulatory requirements. Before use, the informed consent form will be reviewed by the EC. By signing the informed consent form, patients agree to take part in the study.

Confidentiality Policy The investigator will comply with the confidentiality policy as described in the Non- Interventional Trial Agreement.

Study Documents and Case Report Forms The investigator will maintain complete and accurate study documentation in a separate file. Documentation may include medical records, records detailing the progress of the study for each subject, signed informed consent forms, correspondence with the EC, enrollment and screening information, CRFs and laboratory reports. The investigator will comply with the procedures for data recording and reporting.

Document and Data Retention The investigator will retain study documentation and data in accordance with applicable regulatory requirements and the document and data retention policy, as described in the Non-Interventional Study Agreement.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

- Patients with liver cirrhosis of any etiology, diagnosed using imaging and/or histological criteria and observed in the Liver Unit of the "A. Gemelli" University will be included in this study. All patients will sign an informed consent. The severity of liver function failure will be assessed using the Child-Pugh score [11]. Upper gastrointestinal endoscopy will be performed in all patients; the size of esophageal varices will be recorded as well as the presence of previous episodes of gastrointestinal bleeding. All the subjects will be outpatients and the time interval between the follow up visits will be approximately 120 days. The ultrasound criteria for the diagnosis of PVT will be the detection of echogenic material within one or more of the following vessels: portal trunk, right portal branch, left portal branch, splenic vein and superior mesenteric vein. Color and pulsed Doppler analysis will allow to confirm the diagnosis and to distinguish partial from complete obstructive thrombosis and in all cases the Doppler ultrasound diagnosis of PVT will be confirmed by contrast enhanced abdomen computed tomography. The presence and/or extension of the thrombosis to the other major vessels of the portal venous system (mesenteric or splenic vein) will registered in all patients. PVT will be classified according to the extension of thrombosis, as previously reported: grade I is referred to as portal thrombosis confined to the portal vein beyond the confluence of the splenic vein; grade II was a PVT extended to the superior mesenteric vein, but with patent mesenteric vessels; grade III is a PVT extended to the whole splanchnic venous system, but with large collaterals; grade IV is a thrombosis extended to the whole splanchnic venous system with only fine collaterals [12]. All the biochemical and coagulation parameters described below, including ADAMTS-13 and VWF levels, will be measured at each follow up visit.

Exclusion Criteria:

* Exclusion Criteria All patients should not have hepatocellular carcinoma or other malignant tumors, they should not be treated with anticoagulant / antiplatelet agents, not affected by PVT already diagnosed and not suffering from congenital coagulation disorders (haemophilia A / B, von disease Willebrand, another congenital deficiency of coagulation factors) or severe thrombocytopenia (<30,000/µl).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with liver cirrhosis of any etiology, diagnosed using imaging and/or histological criteria and observed in the Liver Unit of the "A. Gemelli" University will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Association of portal vein thrombosis with ADAMTS13 activity | 18 months
  Primary Endpoint To describe in a prospective way the association of both basal ADAMTS-13 level and portal vein flow with development of PVT in cirrhotic patients during 18 months from the enrolment. Measurement of ADAMTS-13 activity. ADAMTS-13 activity was measured in citrated plasma samples by a fluorescence resonance energy transfer (FRET)-based assay,

SECONDARY OUTCOMES:
Analysis of ADAMTS-13 and VWF levels as a function of the etiology of cirrhosis. | 18 months
  The secondary objectives of analyzing the levels of ADAMTS-13 and VWF as a function of the etiology of cirrhosis will be further assessed only after a certified diagnosis of the particular etiologic of cirrhosis. In the case of HCV-associated cirrhosis also the genotype of HCV will be analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Raimondo De Cristofaro, Roma, Italy

REFERENCES:
- [Background] Janssen HL, Meinardi JR, Vleggaar FP, van Uum SH, Haagsma EB, van Der Meer FJ, van Hattum J, Chamuleau RA, Adang RP, Vandenbroucke JP, van Hoek B, Rosendaal FR. Factor V Leiden mutation, prothrombin gene mutation, and deficiencies in coagulation inhibitors associated with Budd-Chiari syndrome and portal vein thrombosis: results of a case-control study. Blood. 2000 Oct 1;96(7):2364-8. PMID 11001884
- [Background] Primignani M, Martinelli I, Bucciarelli P, Battaglioli T, Reati R, Fabris F, Dell'era A, Pappalardo E, Mannucci PM. Risk factors for thrombophilia in extrahepatic portal vein obstruction. Hepatology. 2005 Mar;41(3):603-8. doi: 10.1002/hep.20591. PMID 15726653
- [Background] Parikh S, Shah R, Kapoor P. Portal vein thrombosis. Am J Med. 2010 Feb;123(2):111-9. doi: 10.1016/j.amjmed.2009.05.023. PMID 20103016
- [Background] D'Amico M, Pasta F, Pasta L. Thrombophilic genetic factors PAI-1 4G-4G and MTHFR 677TT as risk factors of alcohol, cryptogenic liver cirrhosis and portal vein thrombosis, in a Caucasian population. Gene. 2015 Aug 15;568(1):85-8. doi: 10.1016/j.gene.2015.05.034. Epub 2015 May 16. PMID 25987440
- [Background] Amitrano L, Guardascione MA, Ames PR, Margaglione M, Iannaccone L, Brancaccio V, Balzano A. Increased plasma prothrombin concentration in cirrhotic patients with portal vein thrombosis and prothrombin G20210A mutation. Thromb Haemost. 2006 Feb;95(2):221-3. doi: 10.1160/TH05-08-0555. PMID 16493481
- [Background] Zoller B, Li X, Sundquist J, Sundquist K. Familial risks of unusual forms of venous thrombosis: a nationwide epidemiological study in Sweden. J Intern Med. 2011 Aug;270(2):158-65. doi: 10.1111/j.1365-2796.2010.02326.x. Epub 2010 Dec 3. PMID 21129048
- [Background] Zocco MA, Di Stasio E, De Cristofaro R, Novi M, Ainora ME, Ponziani F, Riccardi L, Lancellotti S, Santoliquido A, Flore R, Pompili M, Rapaccini GL, Tondi P, Gasbarrini GB, Landolfi R, Gasbarrini A. Thrombotic risk factors in patients with liver cirrhosis: correlation with MELD scoring system and portal vein thrombosis development. J Hepatol. 2009 Oct;51(4):682-9. doi: 10.1016/j.jhep.2009.03.013. Epub 2009 Apr 23. PMID 19464747
- [Background] Ponziani FR, Zocco MA, Campanale C, Rinninella E, Tortora A, Di Maurizio L, Bombardieri G, De Cristofaro R, De Gaetano AM, Landolfi R, Gasbarrini A. Portal vein thrombosis: insight into physiopathology, diagnosis, and treatment. World J Gastroenterol. 2010 Jan 14;16(2):143-55. doi: 10.3748/wjg.v16.i2.143. PMID 20066733
- [Background] Uemura M, Tatsumi K, Matsumoto M, Fujimoto M, Matsuyama T, Ishikawa M, Iwamoto TA, Mori T, Wanaka A, Fukui H, Fujimura Y. Localization of ADAMTS13 to the stellate cells of human liver. Blood. 2005 Aug 1;106(3):922-4. doi: 10.1182/blood-2005-01-0152. Epub 2005 Apr 26. PMID 15855280
- [Background] Lancellotti S, Basso M, Veca V, Sacco M, Riccardi L, Pompili M, De Cristofaro R. Presence of portal vein thrombosis in liver cirrhosis is strongly associated with low levels of ADAMTS-13: a pilot study. Intern Emerg Med. 2016 Oct;11(7):959-67. doi: 10.1007/s11739-016-1467-x. Epub 2016 May 24. PMID 27220954
- [Background] Pugh RN, Murray-Lyon IM, Dawson JL, Pietroni MC, Williams R. Transection of the oesophagus for bleeding oesophageal varices. Br J Surg. 1973 Aug;60(8):646-9. doi: 10.1002/bjs.1800600817. No abstract available. PMID 4541913
- [Background] Yerdel MA, Gunson B, Mirza D, Karayalcin K, Olliff S, Buckels J, Mayer D, McMaster P, Pirenne J. Portal vein thrombosis in adults undergoing liver transplantation: risk factors, screening, management, and outcome. Transplantation. 2000 May 15;69(9):1873-81. doi: 10.1097/00007890-200005150-00023. PMID 10830225
- [Background] Kokame K, Nobe Y, Kokubo Y, Okayama A, Miyata T. FRETS-VWF73, a first fluorogenic substrate for ADAMTS13 assay. Br J Haematol. 2005 Apr;129(1):93-100. doi: 10.1111/j.1365-2141.2005.05420.x. PMID 15801961